CLINICAL TRIAL: NCT04407182
Title: Safety and Efficacy of Viusid and Asbrip in Hospitalized Patients in Teodoro Maldonado Carbo Specialty's Hospital Infected and Diagnosed by SARS-Cov-2 With COVID-19
Brief Title: Safety and Efficacy of Viusid and Asbrip in Hospitalized Patients Infected by SARS-Cov-2 With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IESS-HTMC-JUTD-2020-0305-M
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-05

CONDITIONS: Covid-19; Sars-CoV2; Diabete Mellitus; Cardiopathy; Pulmonary Disease; Renal Disease; Liver Diseases
Keywords: Covid-19; SARS-CoV2; Immuno-modulator; antioxidant; nutritional supplement
MeSH Terms: conditions — COVID-19; Diabetes Mellitus; Heart Diseases; Lung Diseases; Kidney Diseases; Liver Diseases | interventions — Viusid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Viusid Plus Asbrip (Experimental): Patients will be randomized to receive daily doses of 30 ml of Viusid and 10 ml of Asbrip every 8 hours or standard care. Viusid and Asbrip will be administered orally.
  A total of 60 subjects will be randomized 2: 1 in this study. 40 patients will be assigned to Viusid plus Asbrip plus standard of care.
  Treatment duration: 21 days.
  Interventions: Dietary Supplement: Viusid and Asbrip
- Control (No Intervention): A total of 60 subjects will be randomized 2: 1 in this study. 20 Control patients will be assigned to standard of care.
  Treatment duration: 21 days.

INTERVENTIONS:
Dietary Supplement: Viusid and Asbrip — Patients will be randomized to receive daily doses of 30 ml of Viusid and 10 ml of Asbrip every 8 hours plus standard care. Viusid and Asbrip will be administered orally.
  Treatment duration: 21 days.
  Arms: Viusid Plus Asbrip

SUMMARY:
This is a two-arm, open-label, randomized, phase 2, controlled center study to assess the safety and efficacy of Viusid and Asbrip in patients with mild to moderate symptoms of respiratory disease caused by 2019 coronavirus infection.

Patients will be randomized to receive daily doses of 30 ml of Viusid and 10 ml of Asbrip every 8 hours or standard care. Viusid and Asbrip will be administered orally.

A total of 60 subjects will be randomized 2: 1 in this study. 40 patients will be assigned to Viusid plus Asbrip plus standard of care and 20 control patients with standard of care.

Treatment duration: 21 days.

DETAILED DESCRIPTION:
In December 2019, a group of "pneumonia of unknown origin" cases were reported in Wuhan, China. Only a few days later, Chinese health authorities confirmed that this group was associated with the coronavirus and that the disease caused by it was named Coronavirus Disease 2019 (COVID-19) by the WHO. Confirmed by comparative homology analysis, COVID-19 is closely associated with the bat-like severe acute respiratory syndrome (SARS) coronavirus (bat-SL-covzc45 and bat-SL-covzxc21, with 88% identity), but it is a far cry from coronavirus of severe acute respiratory syndrome (SARS-CoV) (about 79%) and coronavirus from respiratory syndrome of the Middle East (MERS-CoV) (about 50%). The National Health Commission of the People's Republic of China reported a total of 77,658 confirmed cases, including 9,162 with serious illnesses and 2,663 deaths as of February 25, 2020.ç

The new pathogen β-coronavirus was initially named as the new coronavirus (2019-nCoV), but on January 12, 2020 the World Health Organization (WHO) named it coronavirus 2019 (COVID-19). Epidemiological reports demonstrated high infectivity from person to person in social, family, and hospital settings. Given this rapid increase in new cases worldwide, the WHO declared a pandemic state 13 The results of a meta-analysis showed that the most prevalent clinical symptom was fever (91.3%, 95% CI: 86-97%), followed by cough (67.7%, 95% CI: 59-76%), fatigue (51.0%, 95% CI: 34-68%) and dyspnea (30.4%, 95% CI: 21-40%). Comorbidities included hypertension, diabetes, respiratory system disease, and cardiovascular disease. For the Chinese Center for Disease Control and Prevention CDC, a suspected or probable case is defined as a case that meets: (1) three clinical criteria or (2) two clinical criteria and one epidemiological criterion. The clinical criteria are: fever; radiographic evidence of pneumonia or acute respiratory distress syndrome; and low or normal white blood cell count or low lymphocyte count. Epidemiological criteria are: living in Wuhan or history of travel to Wuhan within 14 days before the onset of symptoms; contact with patients with fever and symptoms of respiratory infection within 14 days prior to the onset of symptoms; and a link to confirmed cases or groups of suspected cases. Defining a confirmed case, for the first case in a province, is a suspected or probable case with detection of viral nucleic acid at city CDC and provincial CDC. For the second case and all subsequent cases, the definition is a suspected or probable case with detection of nucleic acid from the virus at CDC City. We defined the cases as symptomatic individuals, which could be detected by means of a control temperature across international borders, or who had a disease severity requiring hospital admission, or both, plus travel history to Wuhan. 14 In Ecuador in the city of Guayaquil, the Minister of Health, on February 29, 2020, confirmed the presence of the first "imported" case of Covid-19 in Ecuador. It was an Ecuadorian citizen who arrived from Spain on February 14 at the Guayaquil airport, who had no symptoms. Later days she presented discomfort and fever, reasons for which she was hospitalized and the respective tests were performed for Covid-19 disease, which was positive.

On March 11, 2020, the WHO, the world health organization, officially declares the pandemic caused by the SARS VOC-2 virus and in Ecuador the Emergency Operations Committee is activated, in relation to this committee the following is detailed. The Emergency Operations Committees are components of the Decentralized National Risk Management System, which are responsible for planning and maintaining joint coordination and operation between different levels and functions of the institutions involved in the response and attention to emergencies and disasters in a field territorial defined. On March 12, 2020 two new people tested positive. In total, 19 cases of COVID-19 are registered in Ecuador, the following day the first person died from the coronavirus (COVID-19) occurred in Ecuador. On March 31, 2020, there were 2,240 positive cases for COVID-19, 3,257 suspected, 2,485 discarded from a total of 7,982 samples, 75 confirmed deaths; 61 probable deceased and 54 with hospital discharge. At the beginning of April 2020, the Minister of Public Health, Juan Carlos Zevallos, in a virtual press conference, announced that 100,000 rapid tests and 100,000 PCRs arrived in our country that will serve to expedite the results of the exams for COVID-19.

Until the closing of this project, the records of the MSP indicated that on April 23, 2020, there were 11,183 confirmed cases and 560 people dead. The city of Guayaquil with a population of more than two million inhabitants with the increase in more positive and suspicious cases, became the epicenter of the pandemic at the national level, in this framework, the Teodoro Maldonado Carbo Specialty Hospital located at In the south of the city, it is a third level hospital, since the aforementioned health crisis began with a high influx of patients suspected of covid-19. Current treatment for COVID-19 is supportive, and respiratory failure due to acute respiratory distress syndrome (ARDS) is the leading cause of mortality. Ruan Q et al. Studied the predictors of mortality in a recent retrospective, multicenter study of 150 confirmed cases of COVID-19 in Wuhan, China, including elevated ferritin (mean 1297.6 ng / ml in non-survivors versus 614.0 ng / ml in survivors; p <0 · 001) and IL-6 (p <0 · 0001), suggesting that mortality could be due to viral hyperinflammation. There is an urgent need for effective treatment. The current focus has been on the development of new therapies, which include antivirals and vaccines. Accumulated evidence suggests that a subgroup of patients with severe COVID-19 may have cytokine storm syndrome.

Objectives:

Determine the safety and efficacy of Viusid + Asbrip in hospitalized patients with COVID-19 diagnosis.

Keep security through identification, proper and timely management of adverse events and evaluation of biochemical parameters.

Measure efficacy through clinical improvement: evaluation of radiological signs and blood analysis estableshed in this study.

ELIGIBILITY:
Inclusion Criteria:

* Population over 18 years of age up to 70, sample size 30.
* Subjects with mild to moderate* symptoms of respiratory illness caused by 2019 coronavirus infection as defined below: Mild disease (uncomplicated):
* Diagnosed with COVID-19 by a standardized RT-PCR assay and Mild symptoms, such as fever, runny nose, mild cough, sore throat, malaise, headache, muscle pain, or discomfort, but no shortness of breath and No signs of more serious lower airway disease.
* RR <20, HR <90, oxygen saturation (pulse oximetry)> 93% in ambient air.

  *Moderate illness:
* Diagnosed with COVID-19 by a standardized RT-PCR assay and
* In addition to the above symptoms, more significant lower respiratory symptoms, including difficulty breathing (at rest or with exertion) or
* Signs of moderate pneumonia, including RR ≥ 20 but <30, HR ≥ 90 but less than 125, oxygen saturation (pulse oximetry)> 93% in ambient air, and
* If available, X-ray or computed tomography-based lung infiltrates <50% present 3. 12-lead ECG at rest clinically normal at the screening visit or, if abnormal, not considered clinically significant by the lead investigator.

  4. The subject (or legally authorized representative) provides her informed written consent before starting any study procedure.

  5. Understand and agree to comply with planned study procedures. 6. Women of childbearing potential must agree to use at least one medically accepted method of contraception (eg, barrier contraceptives [condom or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combined oral contraceptives, transdermal patches or rings) ] or intrauterine devices) for the duration of the study.

Exclusion Criteria:

* None

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Symptom resolution | 21 days
  The number of days required to achieve a score of 0 for each symptom category.
  1. Resolution of symptoms: fever (time frame: 21 days) Fever based on a 0-3 scale: 0 = ≤98.6, 1 => 98.6- 100.6, 2 => 100.6 - 102.6, 3 => 102.6
  2. Resolution of symptoms: cough (time frame: 21 days) Cough based on a 0-3 scale: 0 = no cough, 1 = mild, 2 = moderate, 3 = severe
  3. Resolution of symptoms: shortness of breath (time frame: 21 days) Shortness of breath based on a 0-3 scale: 0 = no shortness of breath, 1 = with moderate intensity exercise 2 = walking on a flat surface 3 = shortness of breath when dressing or doing daily activities
  4. Resolution of symptoms: fatigue (period: 21 days) Fatigue based on a 0-3 scale: 1 = mild fatigue, 2 = moderate fatigue, 3 = severe fatigue.
  5. Composite score that includes all symptoms: (time frame: 21 days) Total composite score of symptoms on days 5, 10, 15, and 21 of study supplementation.

SECONDARY OUTCOMES:
Cumulative incidence of disease severity | 21 days
  Disease severity will be measured using a disease severity clinical event scale (assessed until day 21) Change from baseline in the patient's health status on an ordinal scale of 7 categories (time frame: days 3, 7, 14, 21)
  1. death
  2. Hospitalized, with invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, with non-invasive ventilation or high-flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, which does not require supplemental oxygen
  6. Not hospitalized, limitation of activities.
  7. Not hospitalized, without limitations in activities. Note: lower scores mean a worse result.
Complementary drugs required | 21 days
  Differences in the number of patients who received complementary medications for diagnosis between the study arms.
Side effects of supplementation | 21 days
  Differences in the number of patients in the study groups experiencing side effects of the supplements.
Duration of SARS-CoV-2 PCR positivity | 21 days
  PCR analysis at day 0, 7th, 14th and 21th to measure and compare viral load
Concentration of reactive protein c in peripheral blood | 21 days
  Blood biochemical analysis at day 0, 3rd, 7th, 14th and 21th
Incidence of hospitalization | 21 days
  Number of Incidence of hospitalization
Duration (days) of hospitalization | 21 days
  Number of days of hospitalization
Incidence of mechanical ventilation supply | 21 days
  Number of Incidences of mechanical ventilation supply per patient
Duration (days) of mechanical ventilation supply | 21 days
  Number of days with mechanical ventilation supply
Incidence of oxygen use | 21 days
  Number of incidences of oxygen use
Duration (days) of oxygen use | 21 days
  Number of days of oxygen use per patient
Mortality rate | 21 days
  Number of death per group
Time to return to normal activity | 21 days
  Number of days patient need to recover from disease

OTHER OUTCOMES:
Change from baseline in serum cytokine levels | 21 days
  Change from baseline in serum cytokine IL-1 level by blood biochemical analysis at day 0, 3, 7, 14 and 21
Change from baseline in serum cytokine levels | 21 days
  Change from baseline in serum cytokine IL-6 level by blood biochemical analysis at day 0, 3, 7, 14 and 21
Change from baseline in serum cytokine levels | 21 days
  Change from baseline in serum cytokine TNF-α level by blood biochemical analysis at day 0, 3, 7, 14 and 21
Change from baseline in CCR5 receptor occupancy levels for Tregs and macrophages | 21 days
  Change from baseline in CCR5 receptor occupancy levels for Tregs and macrophages by blood biochemical analysis at day 0, 3, 7, 14 and 21
Change from baseline in CD3 +, CD4 + and CD8 + T cell counts | 21 days
  Change from baseline in CD3 +, CD4 + and CD8 + T cell counts by blood biochemical analysis at day 0, 3, 7, 14 and 21.
Change in liver function test | 21 days
  Change in liver function test (AST, ALT and TBIL) by blood biochemical analysis at day 0, 4, 7, 14 and 21.
Change in kidney function test | 21 days
  Change in kidney function with eGFR rate by blood and urinary biochemical analysis at day 0, 4, 7, 14 and 21.
Change in kidney function test | 21 days
  Change in kidney function with creatine clearance rate by blood and urinary biochemical analysis at day 0, 4, 7, 14 and 21.
Change in routine blood test | 21 days
  Change in routine blood test red blood cells concentration by blood biochemical analysis at day 0, 4, 7, 14 and 21.
Change in routine blood test | 21 days
  Change in routine blood test white blood cell concentration by blood biochemical analysis at day 0, 4, 7, 14 and 21.
Change in routine blood test | 21 days
  Change in routine blood test D-dimer level by blood biochemical analysis at day 0, 4, 7, 14 and 21.
Change in routine blood test | 21 days
  Change in routine blood test fibrinogen level by blood biochemical analysis at day 0, 4, 7, 14 and 21.
Change in myocardial enzymes | 21 days
  Change in myocardial enzyme CPK-MB by blood biochemical analysis at daty 0, 4, 7, 14 and 21
Change in myocardial enzymes | 21 days
  Change in myocardial enzymes troponins by blood biochemical analysis at daty 0, 4, 7, 14 and 21

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Especialidades Dr. Teodoro Maldonado Carbo, Guayaquil, Ecuador

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Hui DS, I Azhar E, Madani TA, Ntoumi F, Kock R, Dar O, Ippolito G, Mchugh TD, Memish ZA, Drosten C, Zumla A, Petersen E. The continuing 2019-nCoV epidemic threat of novel coronaviruses to global health - The latest 2019 novel coronavirus outbreak in Wuhan, China. Int J Infect Dis. 2020 Feb;91:264-266. doi: 10.1016/j.ijid.2020.01.009. Epub 2020 Jan 14. No abstract available. PMID 31953166
- [Background] Lu R, Zhao X, Li J, Niu P, Yang B, Wu H, Wang W, Song H, Huang B, Zhu N, Bi Y, Ma X, Zhan F, Wang L, Hu T, Zhou H, Hu Z, Zhou W, Zhao L, Chen J, Meng Y, Wang J, Lin Y, Yuan J, Xie Z, Ma J, Liu WJ, Wang D, Xu W, Holmes EC, Gao GF, Wu G, Chen W, Shi W, Tan W. Genomic characterisation and epidemiology of 2019 novel coronavirus: implications for virus origins and receptor binding. Lancet. 2020 Feb 22;395(10224):565-574. doi: 10.1016/S0140-6736(20)30251-8. Epub 2020 Jan 30. PMID 32007145
- [Background] Yang J, Zheng Y, Gou X, Pu K, Chen Z, Guo Q, Ji R, Wang H, Wang Y, Zhou Y. Prevalence of comorbidities and its effects in patients infected with SARS-CoV-2: a systematic review and meta-analysis. Int J Infect Dis. 2020 May;94:91-95. doi: 10.1016/j.ijid.2020.03.017. Epub 2020 Mar 12. PMID 32173574
- [Background] Rothan HA, Byrareddy SN. The epidemiology and pathogenesis of coronavirus disease (COVID-19) outbreak. J Autoimmun. 2020 May;109:102433. doi: 10.1016/j.jaut.2020.102433. Epub 2020 Feb 26. PMID 32113704
- [Background] Wu JT, Leung K, Leung GM. Nowcasting and forecasting the potential domestic and international spread of the 2019-nCoV outbreak originating in Wuhan, China: a modelling study. Lancet. 2020 Feb 29;395(10225):689-697. doi: 10.1016/S0140-6736(20)30260-9. Epub 2020 Jan 31. PMID 32014114
- [Background] Spina S, Marrazzo F, Migliari M, Stucchi R, Sforza A, Fumagalli R. The response of Milan's Emergency Medical System to the COVID-19 outbreak in Italy. Lancet. 2020 Mar 14;395(10227):e49-e50. doi: 10.1016/S0140-6736(20)30493-1. Epub 2020 Feb 28. No abstract available. PMID 32119824
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- See also: Related Info — https://www.salud.gob.ec/el-ministerio-de-salud-publica-del-ecuador-msp-informa-situacion-coronavirus/
- See also: Related Info — http://www.salud.gob.ec/ecuador-recibio-200-mil-pruebas-para-deteccion-del-covid-19/
- See also: Related Info — https://www.salud.gob.ec/ecuador-registra-2-240-casos-positivos-de-covid-19/
- See also: Related Info — http://www.salud.gob.ec/gobierno-nacional-activado-ante-declaratoria-de-emerge/
- See also: Related Info — http://www.edicionmedica.ec/secciones/salud-publica/primer-caso-de-covid-19-en-ecuador-95377